CLINICAL TRIAL: NCT04816695
Title: Volatolom Variation in Severe COPD During Hospitalization for Exacerbation and After Hospitalization (VOC-BPCO-Exa)
Acronym: VOC-BPCO-Exa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Collaborators: Air Liquide SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020_0005
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation
Keywords: Volatile Organic Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VOC analysis (Experimental): VOC analysis in exhaled air in patients hospitalised for COPD exacerbation
  Interventions: Device: VOC analysis

INTERVENTIONS:
Device: VOC analysis — VOC analysis in exhaled air with e-noses and mass spectrometry.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a public health issue due to its prevalence of 8% in the general population (although it is underestimated), particularly due to the number of severe patients suffering from chronic respiratory failure and the number of hospitalizations estimated at 100,000 each year. Total health insurance expenditure in 2017 for chronic respiratory diseases (excluding cystic fibrosis and cancers) was approximately €3.5 billion, including €1 billion for hospitalizations.

Hospitalizations are mainly related to a worsening of the disease (severe exacerbations mainly of viral and/or bacterial origin). Although the majority of exacerbations are treated on an outpatient basis with antibiotics and/or oral corticosteroids, those occurring in the most severe and often the oldest patients may require hospitalization. It should be noted that almost one out of two patients hospitalized for COPD exacerbation is re-hospitalized within six months; on the other hand, age and length of stay are the two main factors of mortality in the year following hospitalization for COPD in the Intensive Care Unit. Early detection of a worsening of the health status related to COPD could allow appropriate management and avoid at least part of the hospitalizations for exacerbation with a consequent reduction of the associated morbi-mortality.

The objective of this clinical study is to determine the evolution of the profile of volatile organic compounds (VOCs) present in the exhaled air (volatolom) in patients with severe COPD after hospitalization for exacerbation. This step should allow the identification of VOCs (modification of the volatolom) which would be associated with a severe COPD exacerbation, by comparing the volatolom at the acute phase of the exacerbation to the volatoloms during the progressive return to a stable state after hospitalization and to those of patients with a stabilized severe COPD (VOC-BPCO clinical study also sponsored by Foch Hospital)

DETAILED DESCRIPTION:
Patients with severe COPD hospitalized for severe exacerbation (40 patients, ex-smokers or smokers) will be eligible for inclusion in the study.

It is planned to participate in 4 sessions (V1 to V4) of 45 minutes duration for V1 and 30 minutes maximum for V2 to V4, separated by 4 to 6 weeks. All sessions will be carried out in the Pneumology Department of the Foch Hospital, volatolomics platform (Exhalomics®).

Exhalation collection will be performed at each visit in order to perform the volatolom analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe COPD (FEV ≤ 50% of theoretical values) hospitalized for exacerbation;
* COPD treated for at least one year with one (or more successive) combination of at least two inhaled drugs: either a Long-Acting Beta2-Adrenergic bronchodilator (LABA) combined with a corticosteroid (CSI), or a LABA combined with a long-acting anti-cholinergic bronchodilator (LAMA), or a triple combination LABA/LAMA/CSI;
* History of at least one severe COPD exacerbation (treated with antibiotics and/or oral corticosteroids) in the two years preceding the study;
* Ex-smokers (at least 6 months of withdrawal) or active daily smokers of more than 10 pack-years;
* Severe dyspnea in basal state before hospitalization (mMRC stage ≥ 2);
* Age between 40 and 85 years old;
* Perfect understanding of the French language;
* Have signed a consent form;
* Be affiliated to a health insurance plan.

Exclusion Criteria:

* Re-hospitalization for severe exacerbation in the 6 months preceding the study;
* Chronic inflammatory disease (rheumatic, etc...) treated with systemic corticosteroid therapy;
* Long-term oxygen therapy (exclusive ambulatory oxygen therapy is not a non-inclusion criterion);
* Unstable cardiovascular pathology (right or left heart failure, coronary artery disease);
* Cancer under treatment or follow-up;
* Pregnant women;
* Deprived of liberty or under guardianship.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Volatolom variations analysis by mass spectrometry | 4 months
  Analysis of the volatolom by mass spectrometry under quiet breathing conditions during hospitalization for COPD exacerbation and during three successive visits, 4 to 6 weeks apart following hospitalization, upon gradual return to steady state.
Volatolom variations analysis by electronic noses | 4 months
  Analysis of the volatolom by electronic noses under quiet breathing conditions during hospitalization for COPD exacerbation and during three successive visits, 4 to 6 weeks apart following hospitalization, upon gradual return to steady state.

SECONDARY OUTCOMES:
Differences in the profiles of VOCs in the exhaled air according to the treatment of the exacerbation | 4 months
  Analyze the differences in the profiles of VOCs in the exhaled air according to the treatment of the exacerbation (with or without antibiotic/ oral corticosteroid therapy, other criteria: ICU, non-invasive ventilation,...)
Differences in the profiles of VOCs in exhaled air according to smoking habits | 4 months
  Analyze the differences in the profiles of VOCs in exhaled air according to smoking habits (ex-smokers versus active smokers),
Compare VOC profiles to those of patients with severe COPD in a stable state | 4 months
  Comparison of VOC profiles determined from severe COPD patients included in the study versus VOC profiles of stable COPD patients who participated in the VOC-BPCO study (Sponsored by Foch Hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Devillier, PhD, Principal Investigator — Hopital Foch
Locations (1):
- Foch hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: No